CLINICAL TRIAL: NCT05029336
Title: Autologous Hematopoietic Stem Cell Transplant for Children and Young Adults With Life Threatening Autoimmune Diseases
Brief Title: Autologous Stem Cell Transplant (ASCT) for Autoimmune Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Director of Cancer Immunotherapy Program, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-016604
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: open label single arm pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD3/CD19 depleted ASCT (Experimental): The test article is autologous stem cell transplant with a CD3/CD19-depleted stem cell product.
  Interventions: Biological: Depletion of CD3/CD19 in an autologous stem cell transplant

INTERVENTIONS:
Biological: Depletion of CD3/CD19 in an autologous stem cell transplant — The purpose of this study is to determine the safety and feasibility of CD3/CD19 depleted autologous stem cell transplant for the treatment of life threatening autoimmune disease. We will perform CD3/CD19 depletion using the CliniMACs device as a means of purging autoreactive T and B cells from the transfused autologous stem cell product, while retaining some immune function, namely natural killer cells and monocytes in the product.
  Other Names: CD3/CD19 depletion using cliniMACs device

SUMMARY:
A subset of autoimmune diseases (ADs) in children and young adults are life-threatening and unresponsive to conventional treatments. In these patients, the delivery of high dose immunosuppressive therapy followed by autologous stem cell transplant (ASCT) offers a treatment strategy capable of purging the pathogenic, autoreactive immune system and an opportunity for "immune reset." This strategy has been used in adults across a myriad of indications with evidence for efficacy. This study proposes a pilot study to evaluate this therapeutic strategy in children and young adults with systemic sclerosis (SSc) and systemic lupus erythematosis (SLE), two potentially life threatening autoimmune diseases that may response to this therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 ≤ 25 years at time of enrollment.
2. Severe systemic sclerosis or systemic lupus erythematosus based on specific criteria
3. Adequate organ function status
4. No active, untreated infections.

Exclusion Criteria:

1. Previous hematopoietic stem cell transplant (HSCT) or solid organ transplant
2. Pregnancy
3. Ongoing participation in a clinical trial testing an investigational drug or ongoing receipt of disallowed disease modifying anti-rheumatic drugs (DMARD)
4. Severe comorbidity that jeopardizes the ability of the subject to tolerate therapy

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Two-year progression free survival | 2 years
  Survival without evidence of relapse or disease progression

SECONDARY OUTCOMES:
Disease-specific response/progression endpoints: SSc cohort | 24 months following transplant
  o Pulmonary function: Change in forced vital capacity (FVC), total lung capacity (TLC) or diffusing capacity of the lung for carbon monoxide (DLCO) > 10%
Disease-specific response/progression endpoints: SSc cohort | 24 months following transplant
  o Skin condition: An improvement is indicated by a decrease on modified Rodan Skin Score (mRSS) of > 5 points
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 24 months following transplant
  o Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) < 4
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 24 months following transplant
  o Complete remission off therapy (BILAG D/E only or SLEDAI=0 and no SLE treatment except hydroxychloroquine)
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 24 months following transplant
  o Serologic response: presence of positive ANA, anti-dsDNA and anticardiolpin antibody titers
Disease-specific response/progression endpoints: Systemic Lupus Erythematosus (SLE) cohort | 24 months following transplant
  o Serologic response: abnormal complement C3 and C4 levels
Overall survival (OS) | 2 and 5 years following transplant
  Overall survival will be considered as time from transplant to death from any cause
Event free survival (EFS) | 2 and 5 years following transplant
  Events include death, and significant persistent organ damage
  o An event based on organ dysfunction must be documented on at least two occasions, at least three months apart and include: respiratory failure (resting O2 saturation < 88%), renal failure (chronic dialysis) and cardiomyopathy (clinical congestive heart failure New York Class III or IV, left ventricular ejection fraction (LVEF) < 30% by echocardiogram despite therapy)
100 day treatment-related mortality | 100 days from stem cell infusion
  Defined as death from non-disease related causes in the 100 days from stem cell infusion
Time to engraftment | 3 days
  • Achieving an absolute neutrophil count (ANC) > 500 cells/uL and an unsupported platelet count of > 20,000 cells/uL for three consecutive days
Change in quality of life | prior to autologous stem cell transplant (ASCT) until 5 years post-transplant
  * Quality of life will be measured based on the Patient-Reported Outcomes measurement Information System (PROMIS) that evaluates physical, mental and social health in adults and children.
  * patient reported outcome measurement information system (PROMIS) will be administered to each patient (or proxy) prior to autologous stem cell transplant (ASCT) and three times/year for the first two years post-transplant and then annually until five years post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Elgarten, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No